CLINICAL TRIAL: NCT02561325
Title: Comparative Evaluation of the Effect on Blood Pressure of an Equivalent Content of Sodium in the Form of Bicarbonate of Sodium and in the Form of Sodium Chloride, on "Sensitive Sodium" Subjects
Acronym: SODIVASC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CHU-0244
Record Dates: First submitted 2015-09-08; First posted 2015-09-28 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Healthy
Keywords: Blood pressure; Sodium Chloride; Sodium Bicarbonate
MeSH Terms: interventions — Sodium Bicarbonate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- NaCI group (Experimental): a clinical trial protocol intended to highlight a possible differential effect in the biological effects of the same sodium intake (2.56 g / day) orally, depending on the nature salt.
  Interventions: Drug: Sodium Bicarbonate and Sodium chloride
- placebo NaCI (Placebo Comparator): a clinical trial protocol intended to highlight a possible differential effect in the biological effects of the same sodium intake (2.56 g / day) orally, depending on the nature salt.
  Interventions: Drug: Sodium Bicarbonate and Sodium chloride

INTERVENTIONS:
Drug: Sodium Bicarbonate and Sodium chloride

SUMMARY:
Many large-scale epidemiological studies have established a link between the average consumption of table salt (sodium chloride) and blood pressure. In France a survey conducted in 2001 showed that the average consumption of salt is 9 to 10g per people / day, and health authorities considered it appropriate to reduce consumption about 20%, by limiting contributions of sodium in prepared foods, bread.

In terms of basic and clinical research, the biological effects of sodium chloride dietary intake, have been the subject of numerous studies for several decades. This work showed that all subjects do not react uniformly to sodium chloride flows, determining what the investigators call people "sodium-sensitive". For these people the sodium intake elevated blood pressure, much more marked than in subjects called "sodium-resistant."

"Sodium-sensitive" people represent 10 to 30% of the population. A marked over-representation of this phenotype was observed in patients with hypertension or a family history of hypertension.

In addition, studies conducted in animals and humans indicate that sodium intake has a different impact on biological parameters mentioned above, as is done in the form of chloride salt or bicarbonate of sodium.

Based on these factors, investigators developed a clinical trial protocol intended to highlight a possible differential effect in the biological effects of the same sodium intake (2.56 g / day) orally, depending on the nature salt.

DETAILED DESCRIPTION:
Pre-selection: Clinical Pharmacology Center or Cardiology department

Selection - Visit 1 : General practitioner's office or Clinical Pharmacology Center

* Signature of informed consent form
* Check of eligibility criteria
* Clinical exam
* Blood pressure measure
* Blood sample (for renal biology)
* Collection of concomitant treatments
* Collection of food habits
* Delivery of the dietary instructions and forbidden treatments

Phenotyping period : (192 subjects)

All the 192 subjects will realize the 3 first visits in order to determine if yes or no the subjects are "Sodium sensitive".

Selection - Visit 1 : General practitioner's office or Clinical Pharmacology Center

* Signature of informed consent form
* Check of eligibility criteria
* Clinical exam
* Blood pressure measure
* Blood sample (for renal biology)
* Collection of concomitant treatments
* Collection of food habits
* Delivery of the dietary instructions and forbidden treatments

Visit 2: General practitioner's office or Clinical Pharmacology Center

* Collection of adverse events and concomitant treatment
* Check of biological analysis
* Clinical examination
* Blood pressure measure
* Attribution of treatment for 2 weeks
* Delivery of a diary and of the blood pressure measure device

Visit 3 : General practitioner's office or Clinical Pharmacology Center

* Return of the diary, the blood pressure measure device and the treatment
* Collection of adverse events and concomitant treatment
* Extraction of the data of blood pressure
* Delivery of the urinary bottle for the twenty-four-hour urine analysis before Visit 4

Determination of the subjects " sodium sensitive ". Sodium sensitive subjects will continue the study and non-sodium sensitive subjects will stop the study.

Wash-out period n°1 (2 weeks at least) pursuit of the dietary instructions.

Cross over study - Clinical Pharmacology Center :Center (48 subjects)

All the subjects will realize the 4 visits of the cross over study, and will received Nacl and placebo according to the randomisation plan.

Visit 4 and visit 6 contained the same interventions for the participant (exept the consultation with the dietetician) and visit 5 et 7 are the same regarding the interventions for the participant.

First period

Visit 4 - Day 0 :

* Return of the urinary bottle
* Collection of adverse events and concomitant treatment
* Clinical examination
* Blood pressure measure
* Arterial compliance (non invasive)
* Pregancy test (for women of childbearing age)
* Measure of weight and height
* Impedancemetry
* Blood sample for biological analysis (electrolyte pattern + serum creatinine + Renine + Aldosterone + Angiotensin II and MPE assay)
* Assay of urinary sodium excretion
* Consultation with a dietician.
* Delivery of a diet record , and a booklet to be completed every day of the study period
* Reminder of the use of the blood pressure measure device
* Delivery of the study treatment according to the randomisation plan :

6.51 g of NaCl per day to distribute on the various meals + 1.5 liters of spring water (poor in sodium) to drink each day, Or placebo NaCl every day to distribute on the various meals + 1.5 liters of spring water (with sodium bicarbonate) to drink each day.

Every day during 14 days The first take of treatment will be done on the Clinical Pharmacology Center

- Delivery of the urinary bottle for the twenty-four-hour urine analysis before Visit 5

Visit 5 (Day 14) :

* Return of the urinary bottle, of the empty treatment (to check compliance), of the diet record and of the booklet
* Collection of adverse events and concomitant treatment
* Clinical examination
* Blood pressure measure
* Arterial compliance (non invasive)
* Measure of weight
* Impedancemetry
* Blood sample for biological analysis (electrolyte pattern + serum creatinine + Renine + Aldosterone + Angiotensin II and MPE assay)
* Assay of urinary sodium excretion
* Delivery of the urinary bottle for the twenty-four-hour urine analysis before Visit 6

Wash-out 2 (at least 2 weeks) pursuit of the dietary instructions.

Second study period

Visit 6 (day28) - beginning period 2

Visite 7 (Day42) - end of period 2 and end of study

This second period is the same as the first period, except that the subject will not have the consultation with the dietetician and will receive the other study treatment according to the randomization plan.

Ancillary Study This trial contains an ancillary study of genotypage (optional with specific consent of the subject) with the aim of the confrontation with the phenotyping.

For that purpose, a blood sample will be made in the period of selection on the subject who gives their consent, in the same time of the blood sample for renal biology at visit 1.

These results would allow to identify biomarkers of blood pressure sensibility at the sodium.

ELIGIBILITY:
Inclusion Criteria:

* - Systolic Blood pressure between 130-160 mmHg and/or diastolic 90-100, not treated and/or family history of arterial high blood pressure (Father or Mother),
* Between 18 and 75 years old
* Asymptomatic on the cardiovascular plan,
* Absence of known heart disorder,
* Brachial Perimeter between 22 and 42 cms,
* Creatinine clearance in the standards dating less than 12 months, (glomerular filtration rate > 60 ml / mn / 1.73m²),
* Agreeing to drink some sparkling water during the periods of study,
* Effective method of birth control for women with childbearing potential
* Cooperation and understanding enough to conform to the study obligations
* Voluntary gives written informed consent to participate in the study
* Affiliated at system of French social security
* Inscription or acceptation of inscription in the national register of volunteers involved in trials.

Exclusion Criteria:

* -Treated by corticoids
* Treated by prohibited medications
* Pregnant or breastfeeding
* Treated by anti-hypertensive drug
* History of heart disease or ischemic heart disease
* Lack of sinus rhythm
* Renal insufficiency (glomerular filtration rate > 60 ml / mn / 1.73m ²)
* Uncontrolled hypertension (> 160 / 100mmHg)
* Incompatible comorbidity with the study
* BMI > 35 kg / m2
* Invalidating cognitive disorders
* Anxiety to use the device to measure blood pressure alone at home judged by the investigator
* Diabetes (Type I and II)
* Chronic alcoholism
* Sports judged as intense (more than 3 hours per week of intense sports),
* Participation in another clinical trial, located in exclusion period or received benefits > 4500 euros during 12 months before the beginning of trial,
* Cooperation and understanding that do not allow him to follow the trial,
* Patients with minor or under guardianship.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2015-09; Primary Completion 2017-01 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Average value of the mean blood pressures | during the last 3 days of each of the 2 periods of treatment of 14 days
  Average value of the mean blood pressures, collected with the device Microlife BP A200, in the morning and evening during the last 3 days of each of the 2 periods of treatment of 14 days.

SECONDARY OUTCOMES:
Value of Aortic Systolic Pressure (SP) with device Sphygmocor ®, | during the last 3 days of each of the 2 periods of treatment of 14 days.
Value of Pulse Pressure (PP), with device Sphygmocor ®, | during the last 3 days of each of the 2 periods of treatment of 14 days.
Value of the Increase Index (AIX) with the Sphygmocor ®, | during the last 3 days of each of the 2 periods of treatment of 14 days.
Value of the Pusle Wave Velocity with the Sphygmocor ®, | during the last 3 days of each of the 2 periods of treatment of 14 days.
Biological assay of Renine (pg/ml) | during the last 3 days of each of the 2 periods of treatment of 14 days
Values of fat mass, dry mass and water by impedancemetry. | during the last 3 days of each of the 2 periods of treatment of 14 days
Biological assay Aldostéron (pg/ml) | during the last 3 days of each of the 2 periods of treatment of 14 days
Biological assay Angiotensine II (UECA) | during the last 3 days of each of the 2 periods of treatment of 14 days
Biological Assay of the Endotheliales microparticles (nb/µl) | during the last 3 days of each of the 2 periods of treatment of 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Claude DUBRAY, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France